CLINICAL TRIAL: NCT02042534
Title: Rivaroxaban Versus Warfarin in Acute Ischemic Stroke With Atrial Fibrillation: Acute Stroke With Xarelto to Reduce Intracranial Bleeding, Recurrent Embolic Stroke, and Hospital Stay, Phase 2, Conceptual Multicenter Trial
Brief Title: Rivaroxaban Versus Warfarin in Acute Ischemic Stroke With Atrial Fibrillation
Acronym: TripleAXEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Sun U. Kwon, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMI-2013-1013
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: stroke; TIA
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Stroke | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban group for 1 month : initial 5 days after randomization rivaroxaban 10mg QD will be administered. Rivaroxaban 20mg QD, but 15mg in case of Cr CL will be administered for remaining 25 days.
  Interventions: Drug: Rivaroxaban
- Warfarin (Active Comparator): Patients allocated to warfarin receive warfarin plus aspirin 100mg until INR value exceed 1.7 followed by warfarin monotherapy with target INR value of 2.5 [2.0 - 3.0].
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban group receive oral rivaroxaban 10 mg once daily for 5 consecutive days, followed by 20 mg or 15 mg in patients with a calculated creatinine clearance of 30-49 ml/min.
  The dosage of rivaroxaban is leveraged from results of ROCKET-AF trial, where 20 mg of rivaroxaban was shown to offer balanced efficacy and safety.
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Warfarin — To harmonize the warfarin regimen across the sites, fixed algorithm was used in dose calculation, both loading and maintenance, and age, sex, ethnicity, race, weight, height, smoking history, presence of liver disease, indication, baseline INR, target INR and concomitant medication were considered as cofactors (http://www.warfarindosing.org/Source/InitialDose.aspx). Investigators will manage anticoagulation with warfarin per routine clinical care.
  Arms: Warfarin

SUMMARY:
Rationale Acute ischemic stroke due to atrial fibrillation (AF) carries a high risk for early recurrence. In acute stage, guidelines recommend aspirin, but do not recommend anticoagulation due to the increased risk of intracranial bleeding. Since, aspirin has a limited efficacy of preventing recurrent stroke in AF, expert consensus suggests early anticoagulation in non-severe stroke with AF. The current practice for acute ischemic stroke patients with AF is delayed warfarin administration with aspirin use for non-minor stroke or immediate warfarin administration (sometimes with heparin bridging) for minor stroke. However, conventional anticoagulation with warfarin in acute ischemic stroke with AF has the following limitations: 1) risk of intracranial bleeding particularly in acute stage, 2) delayed action and transient paradoxical thrombogenic tendency due to the inhibition of protein C, resulting in the risk of early recurrent embolic stroke, and 3) prolongation of hospitalization waiting for full anticoagulation. In contrast, as compared to warfarin, rivaroxaban is advantageous for reduced risk of intracranial bleeding and immediate anticoagulation efficacy.

Goal The current trial will examine whether early initiation (within 5 days from stroke onset) of rivaroxaban as compared to conventional warfarin would reduce intracranial bleeding, recurrent embolic stroke, and hospital stay in patients with acute ischemic stroke due to AF.

DETAILED DESCRIPTION:
Primary endpoint: Composite of MRI-defined intracranial bleeding and recurrent ischemic lesion within 1 month after randomization (rivaroxaban vs conventional warfarin)

ELIGIBILITY:
Inclusion Criteria: All of below

* Acute ischemic stroke or TIA presumed to be cardioembolic origin (within 5 days from stroke onset) with mild severity: infarct size on DWI less than 1/3 of MCA territory, 1/2 of ACA territory, 1/2 of PCA territory, and 1/2 of one cerebellar hemisphere
* Atrial fibrillation including paroxysmal atrial fibrillation: atrial fibrillation must be documented by ECG evidence (e.g., 12-lead ECG, rhythm strip, Holter, pacemaker interrogation) within 30 days before randomization. This could be obtained from a notation in the subject's record (e.g., medical chart, hospital discharge summary).
* Age ≥19 years
* Informed consent

Exclusion Criteria: Any of below

* Chronic renal failure (GFR less than 30ml/min) or severe hepatic impairment
* Significant hemorrhagic transformation (parenchymal hematoma type I or II by the ECASS definition)
* Stroke mechanism of presumed small vessel occlusion: single small subcortical infarct in the perforating artery territory
* Large hemispheric or cerebellar infarction; larger than 1/3 of MCA territory, 1/2 of ACA territory, 1/2 of PCA territory, and 1/2 of one cerebellar hemisphere
* Mechanical valve requiring warfarin therapy
* Active internal bleeding
* Prior history of symptomatic intracranial bleeding

  : patients with asymptomatic bleedings or microbleedings on MRI are eligible for inclusion
* Major surgery or major trauma within 30 days that might be associated with increased bleeding risk
* Clinically significant gastrointestinal bleeding within 6 months
* Intravenous tissue plasminogen activator use or mechanical embolectomy within 48 hours plus 'significant hemorrhagic transformation as described above (exclusion criteria 2)' or 'large hemispheric infarction or cerebellar infarction as described above (exclusion criteria 4)'

  : patients achieving successful reperfusion without hemorrhage nor large infarction are eligible for enrollment
* Severe anemia: hemoglobin <10 g/dL
* Bleeding diathesis; thrombocytopenia (<90,000/µL, prolonged PT (INR>1.7)
* Sustained uncontrolled hypertension: SBP >180 mmHg or DBP >100 mmHg
* Severe devastating illness, such terminal cancer, hepatic failure; therefore, the participants have a life expectancy less than 6 months.
* Planned invasive procedure with potential for uncontrolled bleeding, including major surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Uck Kwon, PhD., Principal Investigator — Asan Medical Center; Keun-Sik Hong, PhD, Principal Investigator — InjeUniversityIlsanPaikHospital; Young Jae Kim, PhD, Principal Investigator — Ewha Womans University Mokdong Hospital; Yang Ha Hwang, PhD, Principal Investigator — Kyungpook National University Hospital; Jaekwan Cha, PhD, Principal Investigator — Dong-A University Hospital; Woo-Keun Seo, PhD, Principal Investigator — Korea University Guro Hospital; Eung-Gyu Kim, PhD, Principal Investigator — InjeUniversityBusanPaikHospital; Byung-Woo Yoon, PhD, Principal Investigator — Seoul National University Hospital; Kyung-Ho Yu, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hong KS, Kwon SU, Lee SH, Lee JS, Kim YJ, Song TJ, Kim YD, Park MS, Kim EG, Cha JK, Sung SM, Yoon BW, Bang OY, Seo WK, Hwang YH, Ahn SH, Kang DW, Kang HG, Yu KH; Phase 2 Exploratory Clinical Study to Assess the Effects of Xarelto (Rivaroxaban) Versus Warfarin on Ischemia, Bleeding, and Hospital Stay in Acute Cerebral Infarction Patients With Non-valvular Atrial Fibrillation (Triple AXEL) Study Group. Rivaroxaban vs Warfarin Sodium in the Ultra-Early Period After Atrial Fibrillation-Related Mild Ischemic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2017 Oct 1;74(10):1206-1215. doi: 10.1001/jamaneurol.2017.2161. PMID 28892526
- [Derived] Hong KS, Choi YJ, Kwon SU; Triple AXEL Investigators. Rationale and design of Triple AXEL: trial for early anticoagulation in acute ischemic stroke patients with nonvalvular atrial fibrillation. Int J Stroke. 2015 Jan;10(1):128-33. doi: 10.1111/ijs.12386. Epub 2014 Oct 26. PMID 25346499

RESULTS

PARTICIPANT FLOW:
Groups:
- Rivaroxaban: Rivaroxaban group for 1 month : initial 5 days after randomization rivaroxaban 10mg QD will be administered. Rivaroxaban 20mg QD, but 15mg in case of Cr CL will be administered for remaining 25 days.
  Rivaroxaban: Rivaroxaban group receive oral rivaroxaban 10 mg once daily for 5 consecutive days, followed by 20 mg or 15 mg in patients with a calculated creatinine clearance of 30-49 ml/min.
  The dosage of rivaroxaban is leveraged from results of ROCKET-AF trial, where 20 mg of rivaroxaban was shown to offer balanced efficacy and safety.
Period: Overall Study
Arm/Group | Rivaroxaban | Warfarin
Started | 101 | 94
Completed | 101 | 94
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intention-to-treat analysis : The subject who is measured for the primary end point with IP is administered more than at least once after randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Warfarin | Total
Number analyzed (Participants) | 95 | 88 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (10.1) | 70.6 (10.9) | 70.4 (10.4)
Gender [Count of Participants; unit: Participants]
  Female | 40 | 36 | 76
  Male | 55 | 52 | 107
Body Mass Index [Mean (Standard Deviation); unit: kg/㎡] | 24.4 (3.3) | 23.6 (3.1) | 24.0 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intracranial Bleeding and/or Recurrent Ischemic Lesion as Confirmed by MRI Imaging
Description: Intracranial bleeding: symptomatic hemorrhage confirmed by CT or MRI or asymptomatic hemorrhage on follow-up GRE or SWI imaging at 1 month
  Recurrent ischemic lesion: symptomatic ischemic stroke confirmed by relevant neuroimagings or asymptomatic recurrent ischemic lesion on follow-up or FLAIR imaging at 1 month
Time Frame: 1 month after randomization
Population: * modified Intention to treat: 95 / 88 (Rivaroxaban/Warfarin)
  * Per protocol: 93 / 87 (Rivaroxaban/Warfarin)
  * Safety: 98 / 90 (Rivaroxaban/Warfarin)
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 95 | 88
Participants | 47 | 48

2. Secondary Outcome: The Number of Patients With Intracranial Bleeding
Description: Intracranial bleeding confirmed by relevant neuroimagings
Time Frame: at 1 month
Population: Modified ITT
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 95 | 88
Participants | 30 | 25
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Test type: Superiority or Other; p = 0.6765, Chi-squared

3. Secondary Outcome: The Number of Patients With Recurrent Ischemic Lesion
Description: Recurrent ischemic lesion confirmed by relevant neuroimagings
Time Frame: at 1 month
Population: Modified ITT
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 98 | 88
Participants | 28 | 31
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Test type: Superiority or Other; p = 0.3753, Chi-squared

4. Secondary Outcome: Length of Hospitalization
Description: Time to event will be calculated
Time Frame: at 1month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 94 | 88
days | 4.6 (3.9) | 5.6 (4.3)
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Test type: Superiority or Other; p < .0001, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test

5. Secondary Outcome: Number of Participants With Modified Rankin Score of 0 or 1 at Week 4
Description: modified Rankin Score
  0 : No symptoms at all
  1. : No significant disability despite symptoms; able to carry out all usual duties and activities
  2. : Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. : Moderate disability; requiring some help, but able to walk without assistance
  4. : Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. : Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. : Dead
Time Frame: at 1 month
Population: Modified ITT (mRS 0,1 at Week 4, n(%)
Measure: Number; unit: participants
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 95 | 88
participants | 79 | 64
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Test type: Superiority or Other; p = 0.3301, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Groups:
- Rivaroxaban: Safety population : 98 (patients)
  Rivaroxaban group for 1 month : initial 5 days after randomization rivaroxaban 10mg QD will be administered. Rivaroxaban 20mg QD, but 15mg in case of Cr CL will be administered for remaining 25 days.
  Rivaroxaban: Rivaroxaban group receive oral rivaroxaban 10 mg once daily for 5 consecutive days, followed by 20 mg or 15 mg in patients with a calculated creatinine clearance of 30-49 ml/min.
  The dosage of rivaroxaban is leveraged from results of ROCKET-AF trial, where 20 mg of rivaroxaban was shown to offer balanced efficacy and safety.
- Warfarin: Safety population : 90 (patients)
  Patients allocated to warfarin receive warfarin plus aspirin 100mg until INR value exceed 1.7 followed by warfarin monotherapy with target INR value of 2.5 [2.0 - 3.0].
  Warfarin: To harmonize the warfarin regimen across the sites, fixed algorithm was used in dose calculation, both loading and maintenance, and age, sex, ethnicity, race, weight, height, smoking history, presence of liver disease, indication, baseline INR, target INR and concomitant medication were considered as cofactors (http://www.warfarindosing.org/Source/InitialDose.aspx). Investigators will manage anticoagulation with warfarin per routine clinical care.
Arm/Group | Rivaroxaban | Warfarin
Serious Adverse Events (participants affected / at risk) | 6/98 | 5/90
Other Adverse Events (participants affected / at risk) | 46/98 | 51/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (N=98) | Warfarin (N=90)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Stroke in evolution (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (N=98) | Warfarin (N=90)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 6 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
International normalised ratio increased (Investigations) | 1 (1) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Dizziness (Nervous system disorders) | 3 (3) | 8 (9)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 4 (5) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Others (Social circumstances) | 24 (68) | 12 (103)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No